CLINICAL TRIAL: NCT02241603
Title: Insulin Resistance and Reward Signaling in Obesity
Brief Title: Insulin Resistance and Reward
Acronym: IRRSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CLNB-004-13F
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: Insulin resistance; Consummatory Reward
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study. There is a dietary weight loss intervention aiming for ~5-10% weight loss
Who Masked: Participant
Masking Description: participants are expressly assigned to intervention groups through a non-random method based on metabolic testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight loss (Experimental): Obese Veterans will aim to lose 5-10% body weight
  Interventions: Behavioral: Weight loss
- Baseline comparator (No Intervention): Obese Veterans similar to Aim 1 in BMI, age, gender but not insulin sensitivity will not undergo weight loss

INTERVENTIONS:
Behavioral: Weight loss — Obese Veterans will undergo dietary education for weight loss or weight maintenance
  Arms: Weight loss

SUMMARY:
Obesity is a common problem in the Veteran population as at least 1 in 3 Veterans are obese. When obese people eat food they have less response in areas of the brain that sense pleasure (reward). Decreased pleasure response to food predicts future weight gain. It is not known if this poor brain response is reversible or why obese people's brains respond this way. Insulin in the brain regulates the brain's sensing of pleasure. As people gain weight the function of insulin becomes impaired. The investigators will study if impaired function of insulin is related to a poor brain response to food and if this brain response predicts voluntary intake of food and response to a diet. The investigators will also study if improving the function of insulin with weight loss improves the brain response. These studies will improve the understanding as to why weight loss is difficult and inform us if improving insulin signaling is a potential way to treat obesity.

DETAILED DESCRIPTION:
The current research proposal will investigate the relationship of insulin sensitivity to brain reward signaling. In most obese individuals, insulin signaling is impaired (insulin resistance). Preclinical animal studies suggest that insulin resistance in brain regions important for reward contribute to overeating. This proposal aims to test these hypotheses in humans and to determine if these characteristics are pertinent to clinical outcomes (food intake and weight loss). In humans increased body mass index (BMI) and weight gain occur with decreased food consumption-induced neural activation (consummatory reward) in the caudate of the dorsal striatum. It has been speculated that diminished consummatory reward causes overeating and prevents weight loss, however, this hypothesis has not been directly tested. Further, mechanisms for impaired food consumption-induced neural activation in obesity have not been investigated.

The primary research outcomes of the proposed study are: 1) insulin sensitivity determined by hyperinsulinemic euglycemic clamp, 2) food consumption-induced neural activation as determined by blood-oxygen dependent functional magnetic resonance imaging (BOLD fMRI) scanning, 3) caloric intake at a buffet meal, and 4) weight loss during a weight loss intervention. Based on screening and baseline outcome assessments half of participants will be enrolled in a weight loss intervention and then repeat outcomes measures after intervention. Others will only complete baseline outcome measures. Secondary measures of the study include whole brain activation analyses, neuroendocrine hormone measurement at the time of imaging, psychometric measures including eating behaviors and personality characteristics, and measures of reward sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-60yoa, inclusive.
* BMI 30.0 and 45.0 kg/m2, inclusive.
* Normal visual acuity with correction.
* Able to travel regularly to the St. Louis VA and Washington University for research visits.
* Completed signed informed consent form.

Exclusion Criteria:

* Current or history of significant psychiatric disease, including Binge Eating Disorder (BED).
* Current or history of significant substance abuse or extended use of tobacco.
* Contraindications for MRI (e.g., pregnancy, claustrophobia, pacemaker, circumference > 54 inches, weight > 400 lbs, etc.);
* Significant cardiovascular, pulmonary, renal, liver, neurologic, or metabolic disease.
* Diabetes mellitus.
* Significant anemia.
* Treatment with a medication the affects insulin sensitivity.
* Treatment with centrally acting medications.
* Frequent shift work.
* Significant in-mobility or unable to lay on back still for 1 hour.
* History of bariatric surgery.
* Food allergies/ intolerance that would prevent completing study.
* Symptoms concerning for untreated active mental health disease

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
food consumption-induced neural activation | ~4-9months
  food consumption-induced neural activation as determined by blood-oxygen dependent functional magnetic resonance imaging (BOLD fMRI) scanning

CONTACTS AND LOCATIONS:
Overall Officials: Julia P Dunn, MD, Principal Investigator — St. Louis VA Medical Center John Cochran Division, St. Louis, MO
Locations (1):
- St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunn JP, Lamichhane B, Smith GI, Garner A, Wallendorf M, Hershey T, Klein S. Dorsal striatal response to taste is modified by obesity and insulin resistance. Obesity (Silver Spring). 2023 Aug;31(8):2065-2075. doi: 10.1002/oby.23799. PMID 37475685